CLINICAL TRIAL: NCT05824052
Title: Investigating the Impact of Ex Vivo Ozone Injection on Synovial Fluids in Patients Diagnosed With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar State Hospital (Other Government)
Collaborators: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Mustafa Hüseyin Temel, Research Assistant, Uskudar State Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Ozone1
Record Dates: First submitted 2023-04-08; First posted 2023-04-21 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Knee Osteoarthritis
Keywords: Dose-dependent effect; knee osteoarthritis; ozone therapy; pro-inflammatory cytokines; synovial fluid
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ozone

STUDY DESIGN:
Intervention Model Description: Synovial fluid samples taken from patients will be prepared to form 3 separate groups, one fluid will not be treated, one will be injected with 10 gamma and the other with 30 gamma ozone.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (No Intervention): The synovial fluid taken from the patients and not treated in any way.
- Group 2 (Active Comparator): The synovial fluid taken from the patients and injected 10 gamma ozone.
  Interventions: Other: Ozone injection
- Group 3 (Active Comparator): The synovial fluid taken from the patients and injected 30 gamma ozone.
  Interventions: Other: Ozone injection

INTERVENTIONS:
Other: Ozone injection — Ozone injection is a process where ozone gas is injected into a substance or system for various purposes. Ozone gas (O3) is a highly reactive form of oxygen that can be generated through the use of specialized ozone generators. Ozone injection can be used in a variety of applications, including water treatment, air purification, and medical therapy.
  Arms: Group 2; Group 3

SUMMARY:
The objective of this study is to examine the effect of varying ozone doses on the levels of pro-inflammatory cytokines in synovial fluid collected from individuals with knee osteoarthritis.

DETAILED DESCRIPTION:
In this study, synovial fluid samples will be collected from patients diagnosed with knee osteoarthritis for in vitro studies. The synovial fluid will be collected under sterile conditions by a joint puncture, and ultrasonography will be performed before sample collection. The synovial fluid samples will then be transferred to sterile urine culture tubes, with one containing only synovial fluid and the others containing synovial fluid and ozone gas. Afterward, the synovial fluid samples will be centrifuged, and the upper portion will be stored at -80°C for biochemical analyses. The total protein content will be measured using a commercial kit based on the Bradford method, and the total antioxidant level and Total oxidant levels will be measured using commercially purchased kits according to the manufacturer's instructions. The oxidative stress index will be calculated using the formula (TOS/TAS) and will be normalized to the total protein content measured in the synovial fluid.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with knee osteoarthritis.
* Giving consent to participate in the study.

Exclusion Criteria:

- Not giving consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Protein Determination | 1 day
  The the total protein content in synovial fluid samples will be determined using a commercial kit based on the Bradford method (Coomassie Plus, Protein Assay, Thermofisher Scientific, Massachusetts, USA) and will be measured at 595 nm. A rapid and sensitive method will be used for the quantitation of microgram quantities of protein utilizing the principle of protein-dye binding. The Bradford protein test will be based on the principle that when protein molecules bind to Coomassie dye under acidic conditions, the color will change from brown to blue.
Measurement of Total Antioxidant Level (TAL) | 1 day
  TAL refers to the measurement of the total antioxidant capacity of a substance. This capacity measures a substance's ability to prevent harm from free radicals and reactive oxygen species. Measuring the total antioxidant capacity can be done using different laboratory assays and can be affected by various factors, such as diet, lifestyle, and environment.TAL levels of the samples will be measured using commercially purchased kits according to the manufacturer's instructions (Rel Assay Diagnostics, Mega Tıp, Gaziantep, Turkey).
Measurement of Total Oxidant Level (TOL) | 1 day
  TOL refers to the total amount of oxidizing agents, such as ROS, in a substance or biological sample. Oxidative stress is caused by an imbalance between ROS production and antioxidant defense mechanisms, leading to cellular damage. Various lab assays, detecting biomarkers like MDA or protein carbonyls, can measure TOL, which can help diagnose and monitor diseases associated with oxidative stress, like cardiovascular disease and cancer. TOL levels of the samples will be measured using commercially purchased kits according to the manufacturer's instructions (Rel Assay Diagnostics, Mega Tıp, Gaziantep, Turkey).
Oxidative Stress Index (OSI) | 1 day
  OSI is a calculated value that assesses the balance between oxidative stress and antioxidant defense mechanisms in the body by dividing TOS by TAS. A higher OSI value indicates higher oxidative stress and lower antioxidant defense mechanisms. OSI measurement is helpful for diagnosing and monitoring diseases associated with oxidative stress like cardiovascular disease, diabetes, and cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Ata, M.D., Principal Investigator — Sultan Abdulhamid Han Training and Research Hospital
Locations (1):
- Sağlık Bilimleri Üniversitesi Sultan Abdülhamid Han Eğitim ve Araştırma Hastanesi, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared upon reasonable request by the principal investigator.
Supporting Information: Study Protocol, CSR
Time Frame: 1 year
Access Criteria: Individual participant data (IPD) will be shared upon reasonable request by the principal investigator.